CLINICAL TRIAL: NCT01658033
Title: Phase II Study of Bevacizumab Plus Modified FOLFOX6 Regimen as the Salvage Treatment in Patients With Metastatic Breast Cancer
Brief Title: Bevacizumab Plus Modified FOLFOX6 Regimen as the Salvage Treatment in Metastatic Breast Cancer (MBC) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Associate director of medical oncology department, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fudan BR2012-11
Record Dates: First submitted 2012-07-27; First posted 2012-08-06 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer, Her-2 negative Breast Cancer; Avastin, FOLFOX regimen
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Avastin + mFOLFOX6 (Experimental): Avastin plus FOLFOX6 regimen in the management of her-2 negative breast cancer patients.
  Interventions: Drug: Avastin + mFOLFOX6

INTERVENTIONS:
Drug: Avastin + mFOLFOX6 — mFOLFOX6 regimen, repeated every 2 weeks: Oxaliplatin 85 mg/m2，ivgtt； Leucovorin 400 mg/m2,ivgtt； 5-FU 400 mg/m2，iv，and then 2400 mg/m2，civ46h；
  Avastin: Avastin 5mg/kg q2w or 7.5mg/kg q3w
  Other Names: Avastin; Oxaliplatin; Leucovorin; 5-FU

SUMMARY:
The objective of this phase II study is to evaluate efficacy and safety of avastin plus modified FOLFOX6 regimen in HER-2 negative metastatic breast cancer patients. Fifty-five patients will be enrolled into this study.

DETAILED DESCRIPTION:
Anthracyclines and taxanes are the most frequently used agents for breast cancer,both in adjuvant and in first-line metastatic settings.For the patients who do not respond or relapse early after the administration of a taxane or anthracycline regimen,it is clearly needed to explore new combinations and schedules of drugs.Oxaliplatin has shown very promising activity in MBC either in monotherapy or in combination with 5-fluorouracil(5-FU) with or without leucovorin (LV). Avastin is a target therapy with proven efficacy in the treatment of MBC. Avastin plus FOLFOX regimen showed synergetic effet and been used as the standard trial in metastatic colorectal cancer patients. Based on the above reason, we initiate this phase II study to evaluate efficacy and safety of avastin plus modified FOLFOX6 regimen in HER-2 negative metastatic breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. age>=18years
2. Eastern Cooperative Oncology Group (ECOG) performance status (PS) <=2 and a life expectancy >= 12 weeks;
3. histological-proven, HER-2 negative measurable stage IV disease;
4. exposure to anthracyclines, taxanes either in the neoadjuvant/adjuvant or in the metastatic setting and had documented disease progression after the firstline or secondline treatment
5. Patients previously treated with radiotherapy were eligible for the study, provided that measurable disease existed outside the radiation field.
6. At least 3 weeks from the prior chemotherapy or radiotherapy. At least 2 weeks from the prior endocrine therapy.

Exclusion Criteria:

1. Patients with active infection or other serious underlying medical conditions
2. Patients had prior treatment with 5-FU infusion and/or oxaliplatin therapy
3. Inadequate bone marrow, liver, renal, medullary, and cardiac functions
4. Evidence of spinal cord compression or brain metastasis
5. History of another malignancy within the last five years except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix or a contralateral breast cancer
6. Pregnant or lactating women
7. Serious uncontrolled intercurrent infection
8. History or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding
9. Serious non-bleeding wound, peptic ulcer or bone fracture
10. Prior dihypopyrimidine dehydrogenase deficiency
11. Hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanlised antibodies

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-05; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Progression free survival | response evaluation every two cycles

SECONDARY OUTCOMES:
Number of adverse events | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, PhD, Principal Investigator — Medical Oncology Department; Xichun Hu, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Global cancer statistics, 2002. CA Cancer J Clin. 2005 Mar-Apr;55(2):74-108. doi: 10.3322/canjclin.55.2.74. PMID 15761078
- [Background] Kamby C, Vejborg I, Kristensen B, Olsen LO, Mouridsen HT. Metastatic pattern in recurrent breast cancer. Special reference to intrathoracic recurrences. Cancer. 1988 Nov 15;62(10):2226-33. doi: 10.1002/1097-0142(19881115)62:103.0.co;2-d. PMID 3179937
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Background] Pectasides D, Pectasides M, Farmakis D, Bountouroglou N, Nikolaou M, Koumpou M, Mylonakis N, Kosmas C. Oxaliplatin plus high-dose leucovorin and 5-fluorouracil in pretreated advanced breast cancer: a phase II study. Ann Oncol. 2003 Apr;14(4):537-42. doi: 10.1093/annonc/mdg172. PMID 12649097
- [Derived] Li T, Wang B, Wang Z, Ragaz J, Zhang J, Sun S, Cao J, Lv F, Wang L, Zhang S, Ni C, Wu Z, Xie J, Hu X. Bevacizumab in Combination with Modified FOLFOX6 in Heavily Pretreated Patients with HER2/Neu-Negative Metastatic Breast Cancer: A Phase II Clinical Trial. PLoS One. 2015 Jul 17;10(7):e0133133. doi: 10.1371/journal.pone.0133133. eCollection 2015. PMID 26186012